CLINICAL TRIAL: NCT00891735
Title: A Phase III, Double-masked, Multicenter, Randomized, Active Treatment-controlled Study of the Efficacy and Safety of 0.5 mg and 2.0 mg Ranibizumab Administered Monthly or on an As-needed Basis (PRN) in Patients With Subfoveal Neovascular Age-related Macular Degeneration
Brief Title: A Study of Ranibizumab Administered Monthly or on an As-needed Basis in Patients With Subfoveal Neovascular Age-related Macular Degeneration (HARBOR)
Acronym: HARBOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FVF4579g; GX01511 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-12

CONDITIONS: Age-related Macular Degeneration
Keywords: Lucentis; AMD; Age-related macular degeneration; Subfoveal neovascular age-related macular degeneration; Wet AMD; Macular degeneration; Ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Ranibizumab 0.5 mg monthly (Experimental): Patients received ranibizumab 0.5 mg monthly administered intravitreally for 24 months.
  Interventions: Drug: Ranibizumab
- Ranibizumab 2.0 mg monthly (Experimental): Patients received ranibizumab 2.0 mg monthly administered intravitreally for 24 months.
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.5 mg as-needed (pro re nata [PRN]) (Experimental): Patients received ranibizumab 0.5 mg monthly administered intravitreally for 3 months. Thereafter, patients' visual acuity and eye disease activity were assessed monthly for an additional 21 months. If study defined criteria were met at a monthly assessment, patients received ranibizumab 0.5 mg administered intravitreally.
  Interventions: Drug: Ranibizumab
- Ranibizumab 2.0 mg as-needed (pro re nata [PRN]) (Experimental): Patients received ranibizumab 2.0 mg monthly administered intravitreally for 3 months. Thereafter, patients' visual acuity and eye disease activity were assessed monthly for an additional 21 months. If study defined criteria were met at a monthly assessment, patients received ranibizumab 2.0 mg administered intravitreally.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Sterile solution for intravitreal injection.
  Other Names: Lucentis

SUMMARY:
This is a Phase III, multicenter, randomized, double-masked, dose-comparison study of the efficacy and safety of ranibizumab injection administered intravitreally to patients with choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD). Results are presented for the first 12 months of the study.

ELIGIBILITY:
Inclusion Criteria:

* For sexually active women of childbearing potential, agreement to the use of an appropriate form of contraception (or abstinence) for the duration of the study.

Ocular Inclusion Criteria (Study Eye)

* Best corrected visual acuity (BCVA), using Early Treatment Diabetic Retinopathy Study (ETDRS) charts, of 20/40-20/320 (Snellen equivalent).
* Choroidal neovascularization (CNV) lesions with classic CNV component, occult CNV, or with some classic CNV component were permissible.
* Total area of lesion < 12 disc area or 30.48 mm^2.

Exclusion Criteria:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for age-related macular degeneration (AMD) in the study eye.
* Prior treatment with Visudyne(R), external-beam radiation therapy, or transpupillary thermotherapy (TTT) in the study eye.
* Previous intravitreal drug delivery (eg, intravitreal corticosteroid injection, anti-angiogenic drugs, or device implantation) in the study eye.
* Previous treatment or participation in a clinical trial involving anti-angiogenic drugs (Avastin(R), anecortave acetate, protein kinase C inhibitors, etc), in the non-study eye within 3 months of Day 0 (first day of treatment). The patient may not have received Lucentis(R) or Macugen(R) in the non-study eye within 7 days of Day 0.
* Treatment with Visudyne(R) in the non-study eye < 7 days preceding Day 0.
* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either > 50% of the total area of the lesion or > 1 disc area (2.54 mm^2) in size.
* Subfoveal fibrosis or atrophy in the study eye.
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia.
* Retinal pigment epithelial tear involving the macula in the study eye.
* Any concurrent intraocular condition in the study eye (eg, cataract or diabetic retinopathy) that, in the opinion of the investigator, could either: Require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition; or if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity (BCVA) over the 24-month study period.
* Uncontrolled blood pressure.
* Atrial fibrillation not managed by patient's primary care physician or cardiologist within 3 months of screening visit.
* History of stroke within the last 3 months of screening visit.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications.
* Current treatment for active systemic infection.
* Active malignancy.
* History of allergy to fluorescein, not amenable to treatment.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1097 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (94):
- United States (94):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Campbell, California
  - Chico, California
  - La Jolla, California
  - Los Angeles, California
  - Mountain View, California
  - Oakland, California
  - Palm Desert, California
  - Poway, California
  - Sacramento, California
  - San Francisco, California
  - Santa Ana, California
  - Santa Barbara, California
  - Torrance, California
  - Ventura, California
  - Westlake Village, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Danbury, Connecticut
  - Hamden, Connecticut
  - New Haven, Connecticut
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - ‘Aiea, Hawaii
  - Chicago, Illinois
  - Oak Park, Illinois
  - Indianapolis, Indiana
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Portland, Maine
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Jackson, Michigan
  - Edina, Minnesota
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - New Brunswick, New Jersey
  - Northfield, New Jersey
  - Teaneck, New Jersey
  - Vauxhall, New Jersey
  - Great Neck, New York
  - Lynbrook, New York
  - New York, New York
  - Rochester, New York
  - Shirley, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Camp Hill, Pennsylvania
  - Huntingdon Valley, Pennsylvania
  - Johnstown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Mifflin, Pennsylvania
  - Greenville, South Carolina
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - DeSoto, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Temple, Texas
  - The Woodlands, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Milwaukee, Wisconsin
  - Casper, Wyoming

REFERENCES:
- [Derived] Tong N, Fan W, Su L, Ebraheem A, Uji A, Marion K, Sadda S. RELATIONSHIP BETWEEN OPTICAL COHERENCE TOMOGRAPHY BIOMARKERS AND NUMBER OF INTRAVITREAL RANIBIZUMAB INJECTIONS IN EYES WITH NEOVASCULAR AGE-RELATED MACULAR DEGENERATION IN THE HARBOR STUDY. Retina. 2024 Oct 1;44(10):1696-1703. doi: 10.1097/IAE.0000000000004171. PMID 39287532
- [Derived] Kim S, Stockwell A, Qin H, Gao SS, Sagolla M, Stoilov I, Wuster A, Lai P, Yaspan BL, Jeanne M. Rare CIDEC coding variants enriched in age-related macular degeneration patients with small low-luminance deficit cause lipid droplet and fat storage defects. PLoS One. 2023 Apr 20;18(4):e0280484. doi: 10.1371/journal.pone.0280484. eCollection 2023. PMID 37079518
- [Derived] Adrean SD, Chaili S, Hill L, Amador-Patarroyo MJ. PATTERNS OF SUBRETINAL AND/OR INTRARETINAL FLUID RECURRENCE IN PATIENTS WHO RECEIVED AS-NEEDED RANIBIZUMAB THERAPY IN THE HARBOR TRIAL. Retina. 2023 Apr 1;43(4):624-631. doi: 10.1097/IAE.0000000000003708. Epub 2022 Dec 21. PMID 36729084
- [Derived] Staurenghi G, Cozzi M, Sadda S, Hill L, Gune S. Characteristics that Correlate with Macular Atrophy in Ranibizumab-Treated Patients with Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2023 Apr;7(4):300-306. doi: 10.1016/j.oret.2022.11.002. Epub 2022 Nov 11. PMID 36372347
- [Derived] Lally DR, Hill L, Amador-Patarroyo MJ. Subretinal Fluid Resolution and Visual Acuity in Patients with Neovascular Age-Related Macular Degeneration: A HARBOR Post Hoc Analysis. Ophthalmol Retina. 2022 Nov;6(11):1054-1060. doi: 10.1016/j.oret.2022.05.026. Epub 2022 May 30. PMID 35654363
- [Derived] Sheth V, D'Rozario M, Gune S, Blotner S. Fluctuations in central foveal thickness and association with vision outcomes with anti-VEGF therapy for nAMD: HARBOR post hoc analysis. BMJ Open Ophthalmol. 2022 Mar 9;7(1):e000957. doi: 10.1136/bmjophth-2021-000957. eCollection 2022. PMID 35342822
- [Derived] Freund KB, Staurenghi G, Jung JJ, Zweifel SA, Cozzi M, Hill L, Blotner S, Tsuboi M, Gune S. Macular neovascularization lesion type and vision outcomes in neovascular age-related macular degeneration: post hoc analysis of HARBOR. Graefes Arch Clin Exp Ophthalmol. 2022 Aug;260(8):2437-2447. doi: 10.1007/s00417-022-05586-w. Epub 2022 Mar 3. PMID 35239009
- [Derived] Pawloff M, Bogunovic H, Gruber A, Michl M, Riedl S, Schmidt-Erfurth U. SYSTEMATIC CORRELATION OF CENTRAL SUBFIELD THICKNESS WITH RETINAL FLUID VOLUMES QUANTIFIED BY DEEP LEARNING IN THE MAJOR EXUDATIVE MACULAR DISEASES. Retina. 2022 May 1;42(5):831-841. doi: 10.1097/IAE.0000000000003385. PMID 34934034
- [Derived] Holekamp NM, Sadda S, Sarraf D, Guymer R, Hill L, Blotner S, Spicer G, Gune S. Effect of Residual Retinal Fluid on Visual Function in Ranibizumab-Treated Neovascular Age-Related Macular Degeneration. Am J Ophthalmol. 2022 Jan;233:8-17. doi: 10.1016/j.ajo.2021.06.029. Epub 2021 Jul 18. PMID 34289338
- [Derived] Javaheri M, Hill L, Ghanekar A, Stoilov I. Changes in Treatment-Naive Pigment Epithelial Detachments Associated With the Initial Anti-Vascular Endothelial Growth Factor Injection: A Post Hoc Analysis From the HARBOR Trial. JAMA Ophthalmol. 2021 Feb 1;139(2):219-223. doi: 10.1001/jamaophthalmol.2020.5130. PMID 33331859
- [Derived] Sadda SR, Abdelfattah NS, Lei J, Shi Y, Marion KM, Morgenthien E, Gune S, Balasubramanian S. Spectral-Domain OCT Analysis of Risk Factors for Macular Atrophy Development in the HARBOR Study for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2020 Oct;127(10):1360-1370. doi: 10.1016/j.ophtha.2020.03.031. Epub 2020 Apr 2. PMID 32402555
- [Derived] Khurana RN, Chang L, Day BM, Ghanekar A, Stoilov I. Timing of Peak Vision Gains in Patients with Neovascular Age-Related Macular Degeneration Treated with Ranibizumab. Ophthalmol Retina. 2020 Aug;4(8):760-766. doi: 10.1016/j.oret.2020.02.011. Epub 2020 Feb 27. PMID 32387055
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- [Derived] Khurana RN, Hill L, Ghanekar A, Gune S. Agreement of Spectral-Domain OCT with Fluorescein Leakage in Neovascular Age-Related Macular Degeneration: Post Hoc Analysis of the HARBOR Study. Ophthalmol Retina. 2020 Nov;4(11):1054-1058. doi: 10.1016/j.oret.2020.04.016. Epub 2020 Apr 28. PMID 32353536
- [Derived] Patel Y, Miller DM, Fung AE, Hill LF, Rosenfeld PJ. Are Dilated Fundus Examinations Needed for OCT-Guided Retreatment of Exudative Age-Related Macular Degeneration? Ophthalmol Retina. 2020 Feb;4(2):141-147. doi: 10.1016/j.oret.2019.09.006. Epub 2019 Sep 18. PMID 31735634
- [Derived] Khurana RN, Chang LK, Hill LF, Ghanekar A, Stoilov I. The Value of Prior Response to Anti-Vascular Endothelial Growth Factor for Age-Related Macular Degeneration: A HARBOR Subanalysis. Ophthalmol Retina. 2020 Jan;4(1):13-18. doi: 10.1016/j.oret.2019.06.008. Epub 2019 Jul 5. PMID 31416763
- [Derived] Nassisi M, Lei J, Abdelfattah NS, Karamat A, Balasubramanian S, Fan W, Uji A, Marion KM, Baker K, Huang X, Morgenthien E, Sadda SR. OCT Risk Factors for Development of Late Age-Related Macular Degeneration in the Fellow Eyes of Patients Enrolled in the HARBOR Study. Ophthalmology. 2019 Dec;126(12):1667-1674. doi: 10.1016/j.ophtha.2019.05.016. Epub 2019 May 29. PMID 31281056
- [Derived] Hallak JA, de Sisternes L, Osborne A, Yaspan B, Rubin DL, Leng T. Imaging, Genetic, and Demographic Factors Associated With Conversion to Neovascular Age-Related Macular Degeneration: Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2019 Jul 1;137(7):738-744. doi: 10.1001/jamaophthalmol.2019.0868. PMID 31021381
- [Derived] Sarraf D, London NJ, Khurana RN, Dugel PU, Gune S, Hill L, Tuomi L. Ranibizumab Treatment for Pigment Epithelial Detachment Secondary to Neovascular Age-Related Macular Degeneration: Post Hoc Analysis of the HARBOR Study. Ophthalmology. 2016 Oct;123(10):2213-24. doi: 10.1016/j.ophtha.2016.07.007. Epub 2016 Aug 23. PMID 27566855
- [Derived] Frenkel RE, Shapiro H, Stoilov I. Predicting vision gains with anti-VEGF therapy in neovascular age-related macular degeneration patients by using low-luminance vision. Br J Ophthalmol. 2016 Aug;100(8):1052-7. doi: 10.1136/bjophthalmol-2015-307575. Epub 2015 Nov 5. PMID 26541435
- [Derived] Busbee BG, Ho AC, Brown DM, Heier JS, Suner IJ, Li Z, Rubio RG, Lai P; HARBOR Study Group. Twelve-month efficacy and safety of 0.5 mg or 2.0 mg ranibizumab in patients with subfoveal neovascular age-related macular degeneration. Ophthalmology. 2013 May;120(5):1046-56. doi: 10.1016/j.ophtha.2012.10.014. Epub 2013 Jan 23. PMID 23352196

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab 0.5 mg Monthly: Patients received ranibizumab 0.5 mg monthly administered intravitreally for 12 months.
- Ranibizumab 2.0 mg Monthly: Patients received ranibizumab 2.0 mg monthly administered intravitreally for 12 months.
- Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]): Patients received ranibizumab 0.5 mg monthly administered intravitreally for 3 months. Thereafter, patients' visual acuity and eye disease activity were assessed monthly for an additional 9 months. If study defined criteria were met at a monthly assessment, patients received ranibizumab 0.5 mg administered intravitreally.
- Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN]): Patients received ranibizumab 2.0 mg monthly administered intravitreally for 3 months. Thereafter, patients' visual acuity and eye disease activity were assessed monthly for an additional 9 months. If study defined criteria were met at a monthly assessment, patients received ranibizumab 2.0 mg administered intravitreally.
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Started | 275 | 274 | 275 | 273
Completed | 258 | 258 | 263 | 258
Not Completed | 17 | 16 | 12 | 15
Not completed — Adverse Event | 2 | 0 | 2 | 0
Not completed — Death | 8 | 5 | 4 | 5
Not completed — Lost to Follow-up | 2 | 2 | 2 | 2
Not completed — Physician's decision to withdraw patient | 1 | 0 | 0 | 0
Not completed — Patient's decision to withdraw | 4 | 9 | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN]) | Total
Number analyzed (Participants) | 275 | 274 | 275 | 273 | 1097
Age Continuous [Mean (Standard Deviation); unit: years] | 78.8 (8.4) | 79.3 (8.3) | 78.5 (8.3) | 78.3 (8.3) | 78.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 170 | 163 | 156 | 651
  Male | 113 | 104 | 112 | 117 | 446

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Month 12
Description: BCVA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. A decrease in the BCVA score indicates a worsening of vision. A positive change score indicates improvement.
Time Frame: Baseline to Month 12
Population: Intent-to-treat population: All randomized patients. Missing data were imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
Letters | 10.1 (13.3) | 9.2 (14.6) | 8.2 (13.3) | 8.6 (13.8)

2. Secondary Outcome: Number of Ranibizumab Injections up to But Not Including Month 12
Time Frame: Baseline to Month 12
Population: All treated patients. Observed data were used with no imputation.
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 274 | 274 | 275 | 272
Injections | 11.3 (1.8) | 11.2 (2.1) | 7.7 (2.7) | 6.9 (2.4)

3. Secondary Outcome: Percentage of Patients Who Gained ≥ 15 Letters in Best Corrected Visual Acuity (BCVA) From Baseline at Month 12
Description: BCVA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
Percentage of patients | 34.5 [28.9 to 40.2] | 36.1 [30.4 to 41.8] | 30.2 [24.8 to 35.6] | 33.0 [27.4 to 38.5]

4. Secondary Outcome: Percentage of Patients With a Visual Acuity (VA) Snellen Equivalent of 20/40 or Better at Month 12
Description: VA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart starting at a test distance of 4 meters. An increase in the number of lines read correctly by the patient in the ETDRS chart indicates an improvement of vision. The Snellen equivalent of 20/40 is 14 lines correctly read in the EDTRS chart.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
Percentage of patients | 52.4 [46.5 to 58.3] | 50.0 [44.1 to 55.9] | 46.2 [40.3 to 52.1] | 43.6 [37.7 to 49.5]

5. Secondary Outcome: Percentage of Patients With no Evidence of Fluid From Choroidal Neovascularization (CNV) at Month 12
Description: The presence of fluid from choroidal neovascularization (CNV) was assessed by spectral domain optical coherence tomography (SD-OCT). No evidence of fluid was defined as no subretinal fluid thickness, no cystoid spaces, no intraretinal fluid, no pigment epithelial defect thickness, and average central subfield thickness < 270 µm.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
Percentage of patients | 5.1 [2.5 to 7.7] | 5.8 [3.1 to 8.6] | 2.9 [0.9 to 4.9] | 4.8 [2.2 to 7.3]

6. Secondary Outcome: Change From Baseline in Central Foveal Thickness at Day 7 and Months 1, 2, 3, 4, 6, 9, and 12
Description: Central foveal thickness was assessed by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Baseline to Day 7 and Months 1, 2, 3, 4, 6, 9, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
µm
  Day 7 | -104.9 (130.3) | -84.9 (111.3) | -103.5 (141.3) | -100.6 (123.4)
  Month 1 | -141.5 (137.5) | -128.6 (133.3) | -132.6 (148.2) | -146.0 (144.3)
  Month 2 | -152.5 (142.4) | -140.3 (131.1) | -142.9 (141.6) | -156.9 (145.0)
  Month 3 | -157.0 (143.8) | -147.9 (134.3) | -154.5 (147.9) | -164.9 (144.5)
  Month 4 | -164.0 (146.6) | -151.8 (143.3) | -142.7 (153.6) | -159.7 (148.8)
  Month 6 | -162.0 (150.0) | -149.2 (144.0) | -147.5 (151.9) | -159.1 (149.6)
  Month 9 | -164.5 (151.8) | -153.1 (144.8) | -153.5 (147.1) | -157.8 (155.6)
  Month 12 | -172.0 (150.5) | -163.3 (142.6) | -161.2 (152.3) | -172.4 (148.6)

7. Secondary Outcome: Change From Baseline in Macular Volume at Day 7 and Months 1, 2, 3, 4, 6, 9, and 12
Description: Macular volume was assessed by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Baseline to Day 7 and Months 1, 2, 3, 4, 6, 9, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
mm^3
  Day 7 | -0.79 (0.80) | -0.80 (0.76) | -0.72 (0.87) | -0.81 (0.76)
  Month 1 | -1.26 (1.06) | -1.30 (1.15) | -1.16 (1.03) | -1.38 (1.18)
  Month 2 | -1.34 (1.17) | -1.49 (1.31) | -1.30 (1.13) | -1.47 (1.25)
  Month 3 | -1.42 (1.25) | -1.51 (1.32) | -1.43 (1.33) | -1.55 (1.28)
  Month 4 | -1.42 (1.22) | -1.56 (1.31) | -1.31 (1.24) | -1.48 (1.27)
  Month 6 | -1.47 (1.25) | -1.61 (1.34) | -1.35 (1.33) | -1.48 (1.36)
  Month 9 | -1.55 (1.41) | -1.67 (1.34) | -1.35 (1.31) | -1.48 (1.33)
  Month 12 | -1.54 (1.31) | -1.66 (1.37) | -1.41 (1.36) | -1.49 (1.35)

8. Secondary Outcome: Change From Baseline in the Total Area of Choroidal Neovascularization (CNV) and Choroidal Neovascular Leakage at Month 12
Description: The total area of choroidal neovascularization (CNV) and choroidal neovascular leakage was assessed with fluorescein angiography (FA). Area was measured in disc area units; 1 disc area unit = 2.54 mm^2.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Disc area units
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Number analyzed (Participants) | 275 | 274 | 275 | 273
Disc area units
  Change in the total area of CNV | -2.14 (2.40) | -2.42 (2.38) | -1.74 (2.22) | -1.98 (2.39)
  Change in the total area of CNV leakage | -2.35 (2.39) | -2.63 (2.34) | -2.01 (2.28) | -2.22 (2.48)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from Baseline (first treatment day) through Month 12.
Description: Safety population: All patients who received at least 1 study treatment. Adverse events reported here include ocular adverse events in the study eye and fellow eye, as well as non-ocular adverse events.
Arm/Group | Ranibizumab 0.5 mg Monthly | Ranibizumab 2.0 mg Monthly | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN])
Serious Adverse Events (participants affected / at risk) | 66/274 | 54/274 | 57/275 | 54/272
Other Adverse Events (participants affected / at risk) | 240/274 | 243/274 | 250/275 | 239/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg Monthly (N=274) | Ranibizumab 2.0 mg Monthly (N=274) | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) (N=275) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN]) (N=272)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 4 | 4
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 6 | 1 | 2 | 2
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 5 | 1 | 0 | 3
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 1 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1 | 0 | 0 — Fellow eye
Corneal oedema (Eye disorders) | 0 | 0 | 1 | 0 — Study eye
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0 — Study eye
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 — Study eye
Macular hole (Eye disorders) | 0 | 1 | 0 | 0 — Fellow eye
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0 — Study eye
Retinal haemorrhage (Eye disorders) | 0 | 1 | 1 | 1 — Study eye
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 — Study eye
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0 — Study eye
Visual acuity reduced (Eye disorders) | 0 | 3 | 2 | 0 — Study eye
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 — Study eye
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Large intestinal harmorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 2 | 0
Death (General disorders) | 2 | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Device failure (General disorders) | 0 | 0 | 0 | 1
Medical device complication (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Ulcer haemorrhage (General disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 1 | 0
Breast infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 2 | 0 | 0 | 0 — Study eye
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 5 | 6 | 3
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 3
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural heamatoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 2 | 2
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0
Somatic delusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 2 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Thrombosis prophylaxis (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 0 — Fellow eye
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 — Fellow eye
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg Monthly (N=274) | Ranibizumab 2.0 mg Monthly (N=274) | Ranibizumab 0.5 mg As-needed (Pro re Nata [PRN]) (N=275) | Ranibizumab 2.0 mg As-needed (Pro re Nata [PRN]) (N=272)
Age-related macular degeneration (Eye disorders) | 8 | 15 | 15 | 13 — Fellow eye
Conjunctival haemorrhage (Eye disorders) | 63 | 51 | 48 | 41 — Study eye
Detachment of retinal pigment epithelium (Eye disorders) | 4 | 4 | 17 | 11 — Study eye
Eye pain (Eye disorders) | 15 | 25 | 16 | 23 — Study eye
Macular degeneration (Eye disorders) | 12 | 8 | 18 | 15 — Study eye
Retinal haemorrhage (Eye disorders) | 6 | 7 | 14 | 12 — Study eye
Vitreous detachment (Eye disorders) | 22 | 21 | 16 | 27 — Study eye
Vitreous floaters (Eye disorders) | 26 | 15 | 11 | 17 — Study eye
Nasopharyngitis (Infections and infestations) | 17 | 10 | 17 | 23
Sinusitis (Infections and infestations) | 12 | 7 | 27 | 8
Urinary tract infection (Infections and infestations) | 15 | 14 | 17 | 16
Fall (Injury, poisoning and procedural complications) | 14 | 12 | 8 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 6 | 14
Hypertension (Vascular disorders) | 14 | 20 | 21 | 15
Macular degeneration (Eye disorders) | 14 | 12 | 11 | 14 — Fellow eye
Retinal haemorrhage (Eye disorders) | 12 | 15 | 6 | 12 — Fellow eye
Vitreous detachment (Eye disorders) | 20 | 24 | 17 | 13 — Fellow eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.